CLINICAL TRIAL: NCT03362983
Title: Integrated, Multidisciplinary, Person-centered Care for Patients With Complex Comorbidities: Heart, Kidney and Diabetes - a Randomized Trial
Brief Title: Integrated, Multidisciplinary, Person-centered Care for Patients With Complex Comorbidities: Heart, Kidney and Diabetes
Acronym: CareHND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonas Spaak, Professor, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CareHND
Record Dates: First submitted 2017-06-14; First posted 2017-12-05 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus; Chronic Kidney Diseases; Cardiovascular Diseases; Chronic Disease; Multimorbidity
MeSH Terms: conditions — Diabetes Mellitus; Renal Insufficiency, Chronic; Cardiovascular Diseases; Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care HND Intervention (Experimental): Integrated, multidisciplinary, person centered care at HND-centrum.
  Interventions: Other: CareHND
- Standard care (No Intervention): Standard care at separate specialty clinics and primary care as needed.

INTERVENTIONS:
Other: CareHND — Multidisciplinary, integrated, person-centered care at the integrated HND-clinic
  Arms: Care HND Intervention

SUMMARY:
Patient with complex comorbidities present a growing challenge for health-care providers, that the current system is poorly designed to handle. Concomitant cardiovascular disease, renal dysfunction and diabetes represent almost half of all patients attending cardiac, kidney and diabetes clinics. Patients with all three of these will be randomized to standard care or to a combined, integrated, person-centered, intensified chronic disease management.

DETAILED DESCRIPTION:
Patients with concomitant cardiovascular disease, renal dysfunction and diabetes represent almost half of all patients attending cardiac, kidney and diabetes clinics, and about 15 % suffer all three. This proportion of patients with multiple chronic conditions increase markedly by age. These complicated diseases interact, and treatment of one affect the others. Despite this have a progressive subspecialisation caused cardiologist to treat "only" the heart, nephrologists "only" the kidneys and endocrinologists' "only" diabetes. Studies and guidelines follow the same pattern. At best this require patients to visit specialists in each field; at worst result in redundant examinations, under-diagnosis and under-treatment of comorbidities. From the patient perspective, there is a great need for coordination and improvement of the care, not only to reduce disease progression but also to optimise quality of life.

We aim to study if the treatment and outcome for patients with concomitant cardiovascular disease, renal dysfunction and diabetes can be improved through a new model to deliver healthcare. We have designed an integrated clinic to handle all three conditions at the same visit, with a person-centered team-based approach between patients, nurses and physicians, with bi-weekly therapy conferences by dedicated and educated cardiologists, nephrologists and endocrinologists. At these, optimised care-plans are developed, and at following team-visits and phone contacts, these are implemented.

The intervention will be studied in a randomised controlled trial (CareHND) at HND-centrum, a novel integrated outpatient clinic in Stockholm.

Our main hypothesis is that HND-centra results in better care, from several aspects, at lower overall burden on the health care system.

The CareHND study will randomise an estimated 260 patients to HND-centrum or standard care.

The sample size is based on a power calculation for the combined outcome (Project 1): readmissions for heart failure, death, myocardial infarction, end-stage renal disease or TIA / stroke with 2 years follow up.

For Project 2, 3 and 4 detailed below the sample size will be 131. At 131 patients randomized an interim analysis will also be performed for the main outcome, after which the sample size will be adjusted if needed.

Inclusion criteria - CareHND:

1. - Established cardiovascular disease, and:
2. - Diabetes mellitus type 1 or 2, and:
3. - Established kidney disease (eGFR <60 mL/min/m2 or macroalbuminuria).

Intervention:

Combined (nurses, physicians and paramedics), integrated (nephrology, diabetology and cardiology), person-centered, intensified chronic disease management at an integrated clinic for up to 12 months.

Outcome measures:

Project 1: traditional outcome measures including disease progression. Project 2: perceived quality of care. Project 3: value-based analysis of integrated clinic and health management. Project 4: Comparison between Sweden and Canada.

ELIGIBILITY:
Inclusion Criteria:

1. - Established cardiovascular disease (such as history of myocardial infarction, angina, or heart failure requiring hospitalization, previous stroke or TIA with certain diagnosis, and peripheral vascular disease), as well as:
2. - Diabetes mellitus type 1 or 2 (treated diabetes, or new onset diabetes according to WHO criteria or HbA1C > 48, and symptoms, as well as:
3. - Established kidney disease (eGFR <60 mL/min/m2 calculated with the CKD-EPI formula, or an average of the CKD -EPI and Cystatin-C eGFR, or borderline GFR but concomitant microalbuminuria, or macroalbuminuria, or kidney transplant).

Exclusion Criteria:

1 - Inability to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Disease progression (n=260) | 2 years
  Combined death or readmission due to heart failure, myocardial infarction, PCI/CABG, end stage renal failure, acute renal failure or TIA / stroke.
Patient centered outcome measures (n=131) | 1 year
  Perceived quality of care and patient empowerment assessed by a PROMs (Patient Reported Outcome Measure) questionaire with a sum score.
Quality-of-care outcome measures (n=131) | 1 year
  Combined score of achieved target blood pressure, target HbA1C and target LDL.

SECONDARY OUTCOMES:
Organ damage (n=131) | 1 year
  Decline in eGFR
System biology (n=131) | 1 year
  Changes in markers of disease progression in transcriptomics, proteomics and metabolomics.
Health care structure and utilization (n=131) | 1 year.
  Health care utilization measured by number of outpatient and inpatient contacts
Patient safety (n=131) | 1 year
  Using logged patient safety reports.
Interdisciplinary learning (n=20) | 1 year
  Qualitative analysis of interdisciplinary learning between personnel.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas Spaak, MD, PhD, Principal Investigator — Danderyd University Hospital and Karolinska Institutet
Locations (1):
- HND centrum, Danderyd University Hospital, Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Upon individual application and review as required by Swedish law.

DOCUMENTS (1):
  • Study Protocol (2017-11-28): https://cdn.clinicaltrials.gov/large-docs/83/NCT03362983/Prot_000.pdf